CLINICAL TRIAL: NCT00930852
Title: Migraine, Appetite Behaviour and Obesity: is There a Link?. A Pilot Study of Migraine and Appetite Behaviour in Children.
Brief Title: A Pilot Study of Migraine and Appetite Behaviour in Children
Status: Completed | Type: Observational
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: 09/H1017/51; 09/15/RE
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Migraine Disorders; Obesity
Keywords: Migraine; Children; Primary headache disorders; Appetite; Obesity; Feeding Behavior
MeSH Terms: conditions — Migraine Disorders; Obesity; Headache Disorders, Primary; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether there is an association between migraine in children and certain patterns of appetite or eating behaviour that may lead to later obesity.

DETAILED DESCRIPTION:
Migraine is a chronic neurological disorder characterized by recurrent episodes of headache and associated symptoms. The condition affects approximately 11% of the child population and it can impose considerable burdens on the sufferer either due to the headache itself, or associated co-morbidities such as psychological stress, obesity, sleep problems, etc. Increasing attention is focussing on the shared genetic, environmental and neurobiological mechanisms of migraine co-morbidities to gain further insights into improving outcomes.

We are interested in studying eating behaviours in children with migraine since there is evidence that altered patterns of eating behaviour (and underlying changes in appetite) are seen in migraineurs although not studied systematically. Altered appetite and eating behaviours may be a mechanism for the emerging association between obesity (or degree of adiposity) and migraine severity, detected in both adult and paediatric studies to varying extents. Studying the putative association between migraine, degree of adiposity and patterns of eating behaviour in children may help to tease out causal mechanisms, since both migraine and obesity often evolve over the course of childhood.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between 5 years and 16 years of age.
* Clinical diagnosis of migraine (for cases).
* Controls are recruited from children referred with headache, who do not receive diagnosis of migraine.

Exclusion Criteria:

* Adolescents 17 years or over.
* Secondary migraine-like disorder e.g., post-craniotomy headache.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: New referrals to outpatient general paediatric and paediatric neurology service (both accepting primary care referrals) within a single multispecialty children's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pearson's correlation between PedMIDAS score (measure of migraine severity) and eating behaviour subscale score on the Child Eating Behaviour Questionnaire or Dutch Eating Behaviour Questionnaire.

SECONDARY OUTCOMES:
Regression coefficient of PedMIDAS score or categories of headache frequency on eating behaviour subscale scores, with covariates of Achenbach Child Behavior Checklist score, current BMI, age, sex, length of history of migraine.
Descriptive analysis of type and severity of typical food cravings and dietary habits using the Food Craving Inventory score and a food intake questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ram Kumar, MRCP, Principal Investigator — Alder Hey Children's NHS Foundation Trust
Locations (1):
- Alder Hey Children's Hospital, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Background] Bigal ME, Lipton RB, Holland PR, Goadsby PJ. Obesity, migraine, and chronic migraine: possible mechanisms of interaction. Neurology. 2007 May 22;68(21):1851-61. doi: 10.1212/01.wnl.0000262045.11646.b1. PMID 17515549
- [Background] Carnell S, Wardle J. Appetite and adiposity in children: evidence for a behavioral susceptibility theory of obesity. Am J Clin Nutr. 2008 Jul;88(1):22-9. doi: 10.1093/ajcn/88.1.22. PMID 18614720
- [Background] Pinhas-Hamiel O, Frumin K, Gabis L, Mazor-Aronovich K, Modan-Moses D, Reichman B, Lerner-Geva L. Headaches in overweight children and adolescents referred to a tertiary-care center in Israel. Obesity (Silver Spring). 2008 Mar;16(3):659-63. doi: 10.1038/oby.2007.88. Epub 2008 Jan 17. PMID 18239560